CLINICAL TRIAL: NCT03266081
Title: Improving Epiphora & Ptosis With Bupivacaine
Brief Title: Bupivacaine Epiphora Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Albert Wu, Assistant Professor, Ophthalmology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS#: 14-00614
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Epiphora; Ptosis
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Blepharoptosis | interventions — Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 0.75% bupivacaine (Experimental)
  Interventions: Drug: 0.75% bupivacaine

INTERVENTIONS:
Drug: 0.75% bupivacaine — topical anesthetic

SUMMARY:
The objective of this study is to investigate quantitative improvement in excessive tearing after administration of Bupivacaine, a local anesthetic, into the affected eyelids.

ELIGIBILITY:
Inclusion Criteria:

Patients age 18 and above, patients with unilateral or bilateral excessive tearing.

Exclusion Criteria:

Pregnant females, vulnerable populations, patients with severe hepatic disease, or patients using monoamine oxidase inhibitors or tricyclic antidepressants, which are contraindicated with bupivacaine and norepinephrine combinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Lacrimal Tear Lake at 6 months | measurements at baseline and 6 months
  Measurement of the height (in mm) of the tear film in the lower conjunctival cup de sac, obtained during slit lamp examination of the eye

SECONDARY OUTCOMES:
Change from baseline Lid distraction at 6 months | measurements at baseline and 6 months
  distance (in mm) that the eyelids can be maximally pulled from the globe
Change from baseline Lid snap back at 6 months | measurements at baseline and 6 months
  Amount of time (in sec) it takes for the lids to return to their normal anatomical position after being pulled to their maximum excursion with fingers

CONTACTS AND LOCATIONS:
Overall Officials: Albert Y Wu, MD PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No